CLINICAL TRIAL: NCT06607237
Title: Prospective, Single Arm, Open-label Clinical Investigation on the Evaluation of Safety and Efficacy of DM-28 for Treatment of Moderate to Severe Ocular Dryness
Brief Title: Evaluation of Safety and Efficacy of DM-28 for Treatment of Moderate to Severe Ocular Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus Pharma (Industry)
Collaborators: Eurofins Dermscan Pharmascan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23E2474
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Product (Experimental)
  Interventions: Device: DM-28

INTERVENTIONS:
Device: DM-28 — 1 drop in each eye, 4 to 6 times per day

SUMMARY:
This study is a pilot, exploratory study to check safety and efficacy of DM-28 device, a new medical device intended to treat moderate to severe ocular dryness.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a moderate to severe dry eye syndrome.
* Subject with a score ≥ 23 for the OSDI (Ocular Surface Disease Index).
* Subject with at least one eye with:

  * Global ocular staining (cornea and conjunctiva) ≥4 and ≤9 on the Oxford scale (0 to 15)

AND one of the following criteria:

* Schirmer test ≥ 3 mm/5 min and ≤ 9 mm/5 min OR
* Sum of 3 measurements of Tear film Break-Up Time (TBUT) ≤ 30s.

  * Subject, having given freely and expressly his/her informed consent.
  * Subject who is able to comply with the study requirements, as defined in the present CIP, at the Investigator's appreciation (investigator expertise).
  * Subject being affiliated to a health social security system.
  * Female subjects of childbearing potential should use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study, during all the study and at least 1 month after the study end (subject declaration).

Exclusion Criteria:

* Far best corrected visual acuity (FBCVA) < 1/10 (according to Snellen Chart)
* Subject with severe ocular dryness with one of these conditions (investigator expertise):

  * Eyelid or blinking malfunction
  * Corneal disorders not related to dry eye syndrome
  * Ocular metaplasia
  * Filamentous keratitis
  * Corneal neovascularization
* Subject with severe meibomian gland dysfunction (MGD)
* History of ocular trauma, infection or inflammation, not related to dry eye syndrome within the last 3 months prior to the inclusion
* History of ocular allergy or ocular herpes within the last 12 months.
* Any troubles of the ocular surface not related to dry eye syndrome.
* Subject with hypersensitivity to one of the components of the investigational device.
* Subjects who underwent ocular surgery, including laser surgery, in either eye within the last 6 months.
* Use of the following systemic or ocular treatments: isotretinoïd, cyclosporine, tacrolimus, sirolimus, pimecrolimus, punctual plugs, corticoids or dry eye therapy (intense pulse light, stem cells) during the month preceding the inclusion.
* Subjects who have received ocular therapy (either eye) with any ophthalmic medication, except tear substitutes, within 2 weeks prior to study start or expected to receive ocular therapy during the study.
* Any not stabilized systemic treatment, which can have an effect on performance or safety criteria, at the investigator appreciation.
* Pregnant or nursing woman or planning a pregnancy during the study (subject declaration/ pregnancy test).
* Subject deprived of freedom by administrative or legal decision (subject declaration).
* Subject in a social or health institution (subject declaration).
* Subject who is under guardianship or who is not able to express his/her consent (subject declaration/ investigator expertise).
* Subject being in an exclusion period for a previous study (subject declaration).
* Subject suspected to be non-compliant according to the Investigator's judgment (investigator expertise).
* Subject wearing contact lenses during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse device effects | Day 35
  Adverse device effects will be evaluated via ocular examination and ocular symptoms after instillation reported by the subjects
Cornea and conjunctiva staining (Oxford scale) (performance) | Day 35
  Main change from baseline of cornea and conjunctiva staining (Oxford scale form 0 to 15, 15 meaning a worse outcome) in the worse eye

SECONDARY OUTCOMES:
Far best corrected visual acuity (FBCVA) | Day 35
  Change from baseline of FBCVA
General safety | Day 35
  Collection and description of ocular and systemic Adverse Events
Cornea and conjunctiva staining (Oxford scale) | Day 35
  Main change from baseline of cornea and conjunctiva staining (Oxford scale from 0 to 15, 15 meaning a worse outcome) in the contralateral eye
OSDI (questionnaire) | Day 35
  Main change from baseline of Ocular Surface Disease Index (OSDI) score
Schirmer test | Day 35
  Main change from baseline of Schirmer test result in the worse eye and contralateral eye
Tear-Film Break Up Time (TBUT) | Day 35
  Main change from baseline of Tear-Film Break Up Time (TBUT) in the worse eye and contralateral eye
Conjunctival hyperaemia | Day 35
  Main change from baseline of conjunctival hyperaemia using the McMonnies scale (from 0 to 5, 5 meaning a worse outcome) in the worse eye and contralateral eye
Global performance by the investigator | Day 35
  Global performance assessment by the investigator using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Global performance by the patient | Day 35
  Global performance assessment by the patient using a 4-point scale (Unsatisfactory, Not very satisfactory, Satisfactory, Very satisfactory)
Comfort upon device administration | Day 4, Day 11, Day 18, Day 25, Day 32
  Evaluation of the comfort upon device administration by the patient using a 5-points scale (from very uncomfortable to very comfortable)
Patient satisfaction on device performance | Day 0, Day 7, Day 14, Day 21, Day 28, Day 35
  Evaluation of patient satisfaction on 5 Visual Analogical Scales (VAS) from 0 to 100 and calculation of the total score

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Paw, MD, Principal Investigator — Eurofins Dermscan Poland
Locations (2):
- Poland (2):
  - Eurofins Dermscan Poland, Gdansk
  - Tu sie Leczy, Gdansk

IPD SHARING:
Plan to Share IPD: Undecided
Depending on any journal publication of the results